CLINICAL TRIAL: NCT06533969
Title: Assessment of Neural Signals for the Control of Assistive Devices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Jonathan Jagid, Professor of Neurological Surgery, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20190536
Record Dates: First submitted 2024-07-25; First posted 2024-08-01 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injury (SCI), Initial Encounter
Keywords: Brain Computer Interface; Epidural Spinal Cord Stimulation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain Computer Interface-Epidural Spinal Cord Stimulation (BCI-ESCS) (Experimental): Participants in this group will receive a onetime surgery to have the leads implanted temporarily for ESCS which will be triggered through the BCI system. The BCI-ESCS arms will include Upper limb (UL) therapist-guided training, with triggered through a BCI system during task practice. The BCI system will decode motor intention of Upper limb (UL) tasks from cortical signals recorded using EEG system or using their intracranially implanted devices (e.g., ECoG). Participants will perform UL daily activities (e.g., grasping, reaching) tailored to participants deficits. The therapist will facilitate task practice and progress therapy within and between session.
  Subjects will be involved in the intervention for up to 2 months.
  Interventions: Procedure: Epidural Spinal Cord Stimulation; Device: Electrocorticographic; Device: Electroencephalographic

INTERVENTIONS:
Procedure: Epidural Spinal Cord Stimulation — This will be a one time surgery lasting no more than 2 hours where ESCS electrodes will be connected to an external stimulator approved for human research. Stimulation intensity and parameters will be configured before each session for optimal upper extremity motor function.
  The ESCS approach will include surgical implantation of temporarily placed leads in the cervical epidural space and connection cables tunneled percutaneously through the skin for <30 days
  Other Names: ESCS
Device: Electrocorticographic — Neural activity during upper and/or lower extremity tasks will be recorded to characterize the changes that occur in the signals before, during, and after task performance. Observed characteristics of neural signals that are related to the initiation, continuation, or termination of movement will be used to derive control signals that can trigger or enable assistive devices.
  Other Names: ECoG
Device: Electroencephalographic — Neural activity during upper and/or lower extremity tasks will be recorded to characterize the changes that occur in the signals before, during, and after task performance. Observed characteristics of neural signals that are related to the initiation, continuation, or termination of movement will be used to derive control signals that can trigger or enable assistive devices.
  Other Names: EEG

SUMMARY:
The study will investigate the use of motor intention-based cortical signals to trigger epidural spinal cord stimulation (ESCS) with individuals with SCI. Motor intention of UL tasks will be decoded using brain-computer interface (BCI) system based on cortical signals recorded using an Electroencephalographic (EEG) system or using their intracranially implanted devices Electrocorticographic (ECoG).

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 and older
* Able to sign informed consent
* Not participating in other studies that limit participation
* Chronic (>6 month) traumatic Spinal Cord Injury (SCI) (C4-T1 neurological injury with American Spinal Injury Association Impairment Scale (AIS A-D) with some residual function.

Exclusion Criteria:

* Patients that are pregnant
* Patients under the age of 18
* Patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Hand Motor Function | Baseline, up to 2 months post-implant
  Toronto Rehabilitation Institute Hand Function Test (TRI-HFT): Measured on a scale from 0-133 to assess upper extremity manipulation and grip force at time points before and after implant.
  Higher scores indicate better hand motor function.
Change in Hand Motor Evoked Potential (MEP) | Baseline, up to 2 months post-implant
  Change in Motor Evoked Potential (MEP): MEP evaluates corticospinal excitability (strength of the connections between the brain and the muscles). The excitability is measured as a peak-to-peak amplitude in millivolts (mV).

SECONDARY OUTCOMES:
Change in Graded and Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) | Baseline, up to 2 months post-implant
  Graded and Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP): Standardized test to be measured on a scale from 0-116 through the combination of five subset scores to assess grasping ability at time points before and after implant. A composite score will be obtained for strength, muscle force and tasks.
  Higher scores indicate better hand motor function.
Change in Muscle Coordination Measured by Electromyography (EMG) | Baseline, up to 2 months post-implant
  Functional tasks: Assessments to measure reaching ability and obtain muscle coordination via EMG (millivolts).
Change in Movement Kinematics | Baseline, up to 2 months post-implant
  Kinematics data (motion capture, measured in centimeters) at time points before and after implant.
Change in Muscle Strength | Baseline, up to 2 months post-implant
  Muscle force testing: Assessment of changes in muscle strength from measured in Newtons at time points before and after implant.
Change in Quality of Life | Baseline, up to 2 months post-implant
  Quality of Life using the International Spinal Cord Injury - Quality of Life (ISCI-QOL): ISCI-QOL consists of three single items on satisfaction with life as a whole, physical health, and psychological health using a 0-10 scale where 0=complete dissatisfaction; 10=complete satisfaction.
  A composite score will be obtained for this measure.
Change in Independence Measured by Spinal Cord Independence Measure (SCIM III) | Baseline, up to 2 months post-implant
  Independence as measured by Spinal Cord Independence Measure (SCIM III): SCIM III assesses performance in activities of daily living Scores range from 0-100, where a score of 0 defines total dependence and a score of 100 is indicative of complete independence.
Change in Satisfaction of Life | Baseline, up to 2 months post-implant
  Medical Outcomes Study Short Form 36 (SF-36): Patient-reported outcome measurement for health-related quality of life and activities of daily living scored on a scale of 0 (negative health) to 100 (positive health).
Change in Pain Levels | Baseline, up to 2 months post-implant
  Brief Pain Inventory (BPI): A questionnaire for pain will be assessed on a scale of 0 ("no pain") to 10 ("worst imaginable pain") at different points before and after the implant.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan R Jagid, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Lynn Rehabilitation Center, Miami, Florida
  - The Miami Project to Cure Paralysis, Miami, Florida

IPD SHARING:
Plan to Share IPD: No